CLINICAL TRIAL: NCT04133259
Title: An Exploratory Study to Evaluate The Efficacy And Safety of HLX10, A Humanized Monoclonal Antibody Targeting Programmed Death-1 (PD-1) Protein In Chronic Hepatitis B Patients
Brief Title: Evaluate the Efficacy and Safety of HLX10 in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henlix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10/HBV-01
Record Dates: First submitted 2019-10-01; First posted 2019-10-21 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic; Monoclonal antibody
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Antibodies, Monoclonal, Humanized; Injections; Nucleosides; entecavir; Tenofovir

STUDY DESIGN:
Intervention Model Description: Simon's Two-Stage Optimal design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX10, in patients with CHB (Experimental): HLX10: 1 mg/kg at 0, 4th, 8th week (maximum 3 doses). Concomitant antiviral medications: take Nucleoside/nucleotide analogues (NAs) starting from at least 2 weeks before the first dose of HLX10 until 12 weeks after the last dose of HLX10 infusion.
  Interventions: Drug: Recombinant anti-programmed death-1 (PD-1) humanized monoclonal antibody; Drug: Nucleoside/nucleotide analogues

INTERVENTIONS:
Drug: Recombinant anti-programmed death-1 (PD-1) humanized monoclonal antibody — Treatment of CHB patient with HLX10
  Other Names: HLX10 for Injection; HLX10
Drug: Nucleoside/nucleotide analogues — Treatment NAs for chronic hepatitis B subject to achieve adequate HBV viral suppression
  Other Names: Entecavir; Tenofovir disoproxil fumarate

SUMMARY:
A multiple-center, open-label, Phase II clinical trial to evaluate the safety and the efficacy of HLX10 in chronic hepatitis B patients.

DETAILED DESCRIPTION:
This study is multiple-center, open-label, Phase II clinical trial and uses Simon's Two-Stage Optimal design. Subjects with chronic hepatitis B (CHB) will be enrolled sequentially and receive up to 3 doses of HLX10 at 1 mg/kg for four weeks apart.

First six subjects will be enrolled in the safety run-in period. If there are no serious adverse events noticed in these 6 subjects up to 6 weeks after the last infusion of HLX10, additional 11 subjects will be enrolled. These 17 subjects (6+11) will be evaluated for efficacy. In the second stage of trial, 27 additional subjects will be enrolled. Total 44 subjects [stage I (n=17) + stage II (n= 27) = total (n=44)] will be accrued in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible subjects must be 18 years of age or older or per local regulations and younger than 65 years.
2. Subjects with chronic hepatitis B infection with serum HBsAg level > 100 IU/mL. [Chronic hepatitis B infection/carrier status must be confirmed by at least two laboratory results of persistent hepatitis B virus (HBV) infection (positive HBs antigen or HBV DNA) collected 6 months apart before the first infusion of HLX10.]
3. Achieved viral suppression, defined as: HBV DNA level (checked within 4 weeks before the first dose of HLX10) lower than 2000 IU/mL.
4. Subjects must be either (1) under nucleoside/nucleotide analogues (NAs) therapy and has achieved viral suppression at the time of study entry or (2) who currently are not taking anti-viral NAs but be able and willing to take one of the designated NAs for a duration of 14 to 22 weeks (2 weeks before the first dose of HLX10, up to 8 weeks during treatment, 12 weeks after the last dose of HLX10).
5. HBe antigen (checked within 4 weeks before the first dose of HLX10) must be negative.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 at the time of study entry.
7. Able to provide informed consent.
8. Adequate hematologic functions, as defined by: a normal white blood cell count, a normal absolute neutrophil count; a hemoglobin level ≥ 10 gm/dL and a platelet count ≥ 100,000/mm3.
9. Adequate hepatic function defined by: a normal total bilirubin level, alanine transaminase (ALT) level and a prothrombin time of INR < 1.5 times normal.
10. Adequate renal function, as defined by the creatinine clearance rate ≥ 50 mL/minute calculated using Cockcroft-Gault formula. In subject with extreme body weight (BMI < 18.5 or > 30), estimated glomerular filtration rate (eGFR) > 50 mL/min calculated using Modification of Diet in Renal Disease (MDRD) formula is acceptable.
11. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 50% measured by multigated acquisition (MUGA) scan or cardiac ultrasound.
12. Use of effective contraceptive measures if procreative potential exists .
13. Able to be followed up the procedures as required by the study protocol.

Exclusion Criteria:

1. Concurrent unstable or uncontrolled medical conditions which include either one of the followings:

   * Active systemic infections that necessitate antimicrobial therapy;
   * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg), or poor compliance with anti-hypertensive agents;
   * Acute myocardial infarction within 12 months OR clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (class III or IV of New York Heart Association [NYHA]);
   * Uncontrolled diabetes (HbA1c > 9.5% in past three months) or poor compliance with hypoglycemic agents;
   * The presence of chronically unhealed wound or ulcers;
   * Other chronic diseases, which, in the opinion of the investigator, could compromise safety of the subject or the integrity of study.
2. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. (Subjects with a previous malignancy without history of liver involvement and without evidence of disease for ≥ 3 years can participate).
3. Pregnancy (confirmed by urine beta human chorionic gonadotropin [ßHCG]) or breast-feeding.
4. History of human immunodeficiency virus infection (HIV). All subjects must agree to undergone screening for HIV.
5. Subject who has an active or a documented history of autoimmune disease (must be confirmed by negative antinuclear antibodies (ANA), rheumatic factor (RF) and anti-double stranded DNA level (anti-dsDNA)).
6. Subject who currently has hepatitis C (defined as anti-HCV antibody reactive or detectable HCV RNA > 15 IU/L) or hepatitis D (defined as anti-HDV antibody reactive).
7. Subject who has a history of interstitial lung disease.
8. Have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of autoimmune disease.
9. The subject is the investigator, sub-investigator or any one directly involved in the conduct of the study.
10. Subject has a history or current evidence of any condition or disease that could confound the results of the study or is not the best interest of the subject to participate, in the opinion of Investigator.
11. History of alcoholism OR recreational drug use.
12. Preexisting advanced liver disease and cirrhosis subject: advanced hepatic fibrosis and cirrhosis are defined as Fibroscan ≥ 9.5 Kpa or Acoustic radiation force impulse (ARFI) ≥ 1.81 m/sec or Fibrosis-4 (FIB-4) ≥ 3.25 or METAVIR F ≥ 3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of the subjects who achieve 0.5 log decline in HBsAg log10 IU/mL from baseline | 12 week
  Efficacy of HLX10 for treatment of chronic HBV

SECONDARY OUTCOMES:
The proportion of the subjects who achieve 1 log decline in HBsAg log10 IU/mL from baseline | 24 weeks
  Efficacy of HLX10 for treatment of chronic HBV
The proportion of subjects with chronic hepatitis B that achieve HBsAg seroclearance after receiving treatment with HLX10. | 9 months
  HLX10 for curative treatment of chronic HBV
The proportion of subjects with chronic hepatitis B who suffered from hepatitis flare after receiving HLX10 | 9 months
  Safety of HLX10 in treatment of chronic HBV

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, MD, PhD, Principal Investigator — National Taiwan University Hospital; Cheng-Yuan Peng, MD, PhD, Principal Investigator — China Medical University Hospital; Chia-Yen Dai, MD, PhD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospita, Taipei

IPD SHARING:
Plan to Share IPD: No